CLINICAL TRIAL: NCT01725672
Title: An Open-Label, Randomized, Single Dose, Four-way Crossover, Multi-stage Study to Determine the Comparative Bioavailability of Two Fixed Dose Combination Tablet Formulations, 500 mg or 1000 mg Extended Release Metformin and 1 mg or 2 mg Extended Release Glimepiride, in Healthy Adult Male and Female Subjects in the Fed State
Brief Title: Crossover Study to Evaluate the Comparative Bioavailability of Two Fixed Dose Combination Tablet Formulations of Extended Release Metformin and Extended Release Glimepiride in Health Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to changes in EMA guidelines on modified release dosage forms (Feb 2013; EMA/CHMP/EWP/280/96). The Part B formulation would not meet the new guidelines.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116806
Record Dates: First submitted 2012-11-01; First posted 2012-11-14 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: healthy volunteers; Diabetes mellitus; glimepiride; pharmacokinetics; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin; glimepiride

ARMS (6):
- Part A and B:Arm 1: 500 mg metformin XR / 1 mg glimepiride IR (Active Comparator): In Part A and Part B of the study, subjects will receive single dose oral tablets of 500 mg metformin XR and 1 mg glimepiride IR on Day 1 of the respective period per randomized sequence
  Interventions: Drug: Metformin, 500 mg extended release tablet; Drug: Glimepiride, 1 mg immediate release tablet
- Part A and B:Arm 2: 1000 mg metformin XR / 2 mg glimepiride IR (Active Comparator): In Part A and Part B of the study, subjects will receive single dose oral tablets of 1000 mg metformin XR and 2 mg glimepiride IR on Day 1 of the respective period per randomized sequence
  Interventions: Drug: Metformin, 1000 mg extended release tablet; Drug: Glimepiride, 2 mg immediate release tablet
- Part A:Arm 3: 500 mg metformin XR and 1 mg glimepiride XR (Experimental): In Part A of the study subjects will receive single oral dose of 500 mg metformin XR and 1 mg glimepiride XR (FDC1) film coated tablet containing release controlling polymers on Day 1 of the respective period per randomized sequence
  Interventions: Drug: Metformin, 500 mg and Glimepiride, 1 mg extended release film coated tablet containing release controlling polymers
- Part A:Arm 4: 1000 mg metformin XR and 2 mg glimepiride XR (Experimental): In Part A of the study subjects will receive single oral dose of 1000 mg metformin XR and 2 mg glimepiride XR (FDC1) film coated tablet containing release controlling polymers on Day 1 of the respective period per randomized sequence
  Interventions: Drug: Metformin, 1000 mg and Glimepiride, 2 mg extended release film coated tablet containing release controlling polymers
- Part B:Arm 5: 500 mg metformin XR and 1 mg glimepiride XR (Experimental): In Part B of the study subjects will receive single oral dose of 500 mg metformin XR and 1 mg glimepiride XR (FDC3) tablet coated with release controlling polymers on Day 1 of the respective period per randomized sequence
  Interventions: Drug: Metformin, 500 mg and Glimepiride, 1 mg extended release tablet coated with release controlling polymers
- Part B:Arm 6: 1000 mg metformin XR and 2 mg glimepiride XR (Experimental): In Part B of the study subjects will receive single oral dose of 1000 mg metformin XR and 2 mg glimepiride XR (FDC4) tablet coated with release controlling polymers on Day 1 of the respective period per randomized sequence
  Interventions: Drug: Metformin, 1000 mg and Glimepiride, 2 mg extended release tablet coated with release controlling polymers

INTERVENTIONS:
Drug: Metformin, 500 mg extended release tablet — In Part A and Part B of the study, Metformin 500 mg XR tablet will be administered with 240 millilitre (mL) water ; 125 mL of LUCOZADE was administered every 30 mins for 4 hours after dosing.
  Arms: Part A and B:Arm 1: 500 mg metformin XR / 1 mg glimepiride IR
Drug: Metformin, 1000 mg extended release tablet — In Part A and Part B of the study, Metformin 1000 mg XR tablet will be administered with 240mL water; 125 mL of LUCOZADE was administered every 30 mins for 4 hours after dosing.
  Arms: Part A and B:Arm 2: 1000 mg metformin XR / 2 mg glimepiride IR
Drug: Glimepiride, 1 mg immediate release tablet — In Part A and Part B of the study, Glimepiride 1 mg IR tablet will be administered with 240mL water; 125 mL of LUCOZADE was administered every 30 mins for 4 hours after dosing.
  Arms: Part A and B:Arm 1: 500 mg metformin XR / 1 mg glimepiride IR
Drug: Glimepiride, 2 mg immediate release tablet — In Part A and Part B of the study, Glimepiride 2 mg IR tablet will be administered with 240mL water; 125 mL of LUCOZADE was administered every 30 mins for 4 hours after dosing.
  Arms: Part A and B:Arm 2: 1000 mg metformin XR / 2 mg glimepiride IR
Drug: Metformin, 500 mg and Glimepiride, 1 mg extended release film coated tablet containing release controlling polymers — In Part A of the study, 1 XR film coated tablet combination of Metformin 500 mg and Glimepiride 1 mg will be administered with 240 mL water; 125 mL of LUCOZADE was administered every 30 mins for 4 hours after dosing.
  Arms: Part A:Arm 3: 500 mg metformin XR and 1 mg glimepiride XR
Drug: Metformin, 1000 mg and Glimepiride, 2 mg extended release film coated tablet containing release controlling polymers — In Part A of the study, 1 XR film coated tablet combination of Metformin 1000 mg and Glimepiride 2 mg will be administered with 240 mL water; 125 mL of LUCOZADE was administered every 30 mins for 4 hours after dosing.
  Arms: Part A:Arm 4: 1000 mg metformin XR and 2 mg glimepiride XR
Drug: Metformin, 500 mg and Glimepiride, 1 mg extended release tablet coated with release controlling polymers — In Part B of the study, 1 XR tablet combination of Metformin 500 mg and Glimepiride 1 mg will be administered with 240 mL water; 125 mL of LUCOZADE was administered every 30 mins for 4 hours after dosing.
  Arms: Part B:Arm 5: 500 mg metformin XR and 1 mg glimepiride XR
Drug: Metformin, 1000 mg and Glimepiride, 2 mg extended release tablet coated with release controlling polymers — In Part B of the study, 1 XR tablet combination of Metformin 1000 mg and Glimepiride 2 mg will be administered with 240 mL water; 125 mL of LUCOZADE was administered every 30 mins for 4 hours after dosing.
  Arms: Part B:Arm 6: 1000 mg metformin XR and 2 mg glimepiride XR

SUMMARY:
This is a an open-label, randomized, single dose, four-way crossover, multi-stage study enrolling 20 healthy adult male and female subjects per part. This study consists of two separate parts (Part A and B) with each part comprising four treatment periods. Each subject will participate in all four treatment periods per part; Subjects may not enrol in both Parts A and B.

This study is being conducted to compare the pharmacokinetics (PK) of two extended release fixed dose combinations (FDC) oral formulations of metformin and glimepiride at two doses, 500mg/1mg and 1000mg/2mg, with each FDC formulation to be administered orally as a single dose and compared with the commercially available formulations of metformin extended release (XR) (GLUCOPHAGE ™ Sustained Release [SR]) and glimepiride immediate release (IR) (AMARYL ™).

Part A of study will evaluate the bioavailability of a formulation comprising a film coated tablet containing release controlling polymers; and Part B will evaluate the bioavailability of a formulation comprising a tablet coated with release controlling polymers.

In each part there will be 4 treatment periods. During each period, subjects will be randomized sequentially to receive a single dose of a reference treatment of 500 mg metformin XR / 1 mg glimepiride IR; and a reference treatment of 1000 mg metformin XR / 2 mg glimepiride IR; and an FDC tablet containing 500 mg metformin XR and 1 mg glimepiride XR; and an FDC tablet containing 1000 mg metformin XR and 2 mg glimepiride XR.Serial PK sampling for up to 36 hours and safety assessments will be performed. Each period will be separated by a washout period of at least 5 days and a follow-up visit will occur 14 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between 18 and 65 years of age inclusive with body weight >= 50 kg and body mass index (BMI) within the range 19 to 32 kilogram/meter squared
* Alanine aminotransferase (ALT) alkaline phosphatase and bilirubin <or=1.5x upper limit of normal (ULN).
* Normal ECG measurements. Average QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 millisecond or QTcF <480 msec in subjects with Bundle Branch Block based on an average from three electrocardiograms (ECGs) obtained over a brief recording period.
* Female subjects of non-child bearing potential. Females of child bearing potential are eligible to enter if they are not pregnant and willing to use protocol-specified methods of contraception to prevent pregnancy until 14 days post-last dose of metformin/glimepiride.
* Capable of giving written informed consent

Exclusion Criteria:

* The subject has a positive: drug/alcohol screen, Hepatitis, HIV screen
* Abuse of alcohol
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Exposure to more than four new investigational chemical entities within 12 months prior to the first dosing day
* Participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Donation of more than 500 mL blood within a 56 day period
* Pregnant or lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* Subject having positive urinary cotinine levels indicative of use of tobacco or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose
* Subjects having asthma or are positive carbon monoxide (CO) on admission to the Unit
* Unable to refrain from the use of prescription or non-prescription drugs within 7 days prior to first dose of study medication, unless approved by the Investigator and GSK Medical Monitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2013-08-21 (Actual); Study Completion 2013-08-21 (Actual)

PRIMARY OUTCOMES:
Cmax of metformin | At regular timepoints on Day 1 (0.5, 1, 1.5, ,2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 hours post dose) and once at Day 2 (36 hours post dose) of each of the 4 treatment periods in Part A and Part B
  The PK parameter: maximum concentration (Cmax) will be determines from the plasma concentration-time data. To select the dose of metformin and glimepiride that achieves the best PK profile Cmax will be measured
AUC(0-t) and AUC(0-inf) for metformin and glimepiride | At regular timepoints on Day 1 (0.5, 1, 1.5, ,2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 hours post dose) and once at Day 2 (36 hours post dose) of each of the 4 treatment periods in Part A and Part B
  The PK parameters: Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable AUC(0-t) concentration; and area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time AUC(0-∞) will be determines from the plasma concentration-time data. To select the dose of metformin and glimepiride that achieves the best PK profile AUC(0-t) and AUC(0-∞) will be measured

SECONDARY OUTCOMES:
Tmax and t1/2 of of metformin and glimepiride | At regular timepoints on Day 1 (0.5, 1, 1.5, ,2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 hours post dose) and once at Day 2 (36 hours post dose) of each of the 4 treatment periods in Part A and Part B
  The PK parameters: Time of occurrence of Cmax (tmax); and terminal phase half-life (t½) will be determines from the plasma concentration-time data. To select the dose of metformin and glimepiride that achieves the best PK profile tmax and t1/2 will be measured , as data permit
Percentage AUCex for metformin and glimepiride; and AUC(0-∞), AUC (0-t) for metformin and glimepiride in relevant treatments | At regular timepoints on Day 1 (0.5, 1, 1.5, ,2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 hours post dose) and once at Day 2 (36 hours post dose) of each of the 4 treatment periods in Part A and Part B
  Percentage of AUC(0-∞) obtained by extrapolation (%AUCex), area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-∞)) and area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC (0-t))will be determined from the plasma concentration-time data
Number of subjects with adverse events (AE)s | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 13 weeks
  Comparison of adverse events (as determined by vital signs and electrocardiogram measurements and clinical lab results) after administration of two metformin and glimepiride fixed dose combinations in comparison to reference treatment (to determine the safety and tolerability) in Part A and Part B of the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116806 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116806?search=study&study_ids=116806#rs
- Available data/document: Clinical Study Report: 116806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register